CLINICAL TRIAL: NCT02486172
Title: Development and Evaluation of A Peer Support Program for Type 2 Diabetes Patients in Hong Kong as Quality Improvement in Diabetes Care Service
Brief Title: Multi-centre Peer Support Program in Type 2 Diabetes Patients in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Rebecca Yee-Man Wong, Clinical Tutor (Honorary), Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CRE Ref. No. 2014.513_FR
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes; Peer Group
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peer supporter (Other): Peer support program
  Interventions: Behavioral: Peer support program

INTERVENTIONS:
Behavioral: Peer support program — Peer support program as an additional service to the routine clinical service

SUMMARY:
This is a pre-and-post study with a study duration of one year involving 7 diabetes centres in Hong Kong. A group of motivated patients with type 2 diabetes will be trained as peer supporters in two training workshops. Patients who may benefit from peer support program will be recruited as peers. In the one year study period, peer supporters are required to have 2 face-to-face interviews and 12 phone calls. Clinical parameters and psycho-behavioral parameters of both peer supporters and peers will be evaluated at the baseline and at the end of the study.

DETAILED DESCRIPTION:
Aim of the Study:

1. To evaluate the impact of peer support program on various clinical, psycho-behavioral outcomes and health utilization outcomes in Hong Kong Chinese with type 2 diabetes
2. To evaluate the feasibility of a peer support program in Hong Kong
3. To evaluate the sustainability of a peer support program in Hong Kong

Duration of the program = 12 months

Indicators and targets:

* Number of peer supporters recruited: 12
* Number of peers recruited = 50
* Number of peer supporter training sessions = 2
* Number of reunion sessions for peer supporters with the investigators = 4
* Minimum number of telephone calls made by peer supporter = 12 for each peer

Method:

1. The diabetes nurses from 7 diabetes centres of public hospitals in Hong Kong will recruit peer supporters and peers in the first 3 months of the project.
2. Nurses will compile list of potential patients to invite to become peer supporters.
3. Selected potential peer supporters will attend 2 half-day training sessions by the diabetes nurses and social workers from the Community Rehabilitation Network according to specially-designed curriculum. In sum, it includes revision of diabetes knowledge, self-management, lifestyle modification, debriefing and rapport building skills. Patients will be evaluated at the end of the training course by social workers and nurses to ensure they are ready to be peer supporters.
4. Diabetes nurses will recruit patients as peers when they attend to the diabetes centre for routine diabetes care services such as complication screening, diabetes group education and nurse-led clinics.
5. Each peer supporter will be matched to 5 peers in the beginning. In case when the peer supporter quitted before the study ends, his/her peers will be directed to another peer support group. The maximum number of peers in each support group is 6.
6. A 2-hour face-to-face introduction of the peer supporters and peers will be held at the diabetes centre when the study begins.
7. Peer supporters will be expected to carry out a minimum of12 phone calls over the next 12 months (one call every 2 weeks for 3 months; one call every month for the second 3 months, one call every 2 months for the last 6 months). Calls will be guided by a call checklist. Both peer supporters and peers will be encouraged to call one another ad lib. Peer supporters will return checklists to the program coordinator, recording the frequency, length, and nature of their interactions with peers

   In the first month of the peer support group, social workers from the Community Rehabilitation Network will contact peer leaders by phone to further foster the peer leader to be committed to the program and to increase their confidence in supporting their peers.

   Two large gatherings for all participants will be organized by the investigators at around 4-8 months after the study and near to the study completion.
8. All peer supporters and peers will receive usual medical follow-up at their original clinics.
9. Peer supporters will have reunion workshop at the diabetes centre with the nursing team and social worker every 2 months throughout the intervention. The workshop will last around 1 hour and it will address any issues the peer supporters encounter, provide some educational by a medical professional, and will facilitate sharing amongst peer supporters to develop a peer supporter network.
10. Surveys for peer supporters and involved staff will also be collected during the debriefing sessions to identify difficulties peer supporters are facing and to better inform ongoing training and education. Surveys will also be administered to peers at the end of the study to obtain opinions and suggestions about their peer support experience.
11. The intervention duration will be 12 months. However peers are encouraged to keep regular contact with peer leaders even after the intervention period ends.
12. A focus-group interview will be conducted by a trained psychologist to two of the peer groups to evaluate participants' satisfaction

Progress tracking:

Clinical, behavioral, and psychological data will be collected at baseline and at the end of the study (12 months):

1. Clinical measures to be done in introduction session and in the second large group gathering: Blood pressure Adiposity (body weight, waist circumference and body mass index)
2. Biochemical measures (HbA1c and lipid profile) were retrieved via the hospital Central Computer System within 2 months of the study starting date and the end date
3. Psychological measures, using validated self-administered questionnaires, to be completed in introduction session and in the second large group gathering:

World Health Organization quality of life questionnaire (WHO-QoL-26) for quality of life 15-item Chinese Diabetes Distress Scale (CDDS-15) for diabetes distress 8-item Patient Health Questionnaire for depressive symptoms EQ5D for quality of life Summary of Diabetes Self Care Activities (SDSCA) for adherence to diabetes self-care

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Age between 18-75 years inclusive
3. Chinese ethnicity
4. High risk patients for poor diabetes control based on the self-administered questionnaire designed by the study team

Exclusion Criteria:

Exclusion criteria for peer supporters:

1. Failure to have 100% attendance rate in the peer supporters training program
2. Inadequate knowledge about diabetes after training program as judged by study investigators

Exclusion criteria for the peers:

1. No access to telephone
2. Unable to speak Cantonese
3. Unable to understand the scope of the project
4. Serious mental or physical disability that prevents one from meeting and communicating regularly with peer supporter
5. Serious medical illness with expected life expectancy < 1 years such as terminal cancer
6. Participation in any diabetes quality improvement program in the past 2 years such as peer support program, Joint Asia Diabetes Evaluation Program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Glycaemic control | 12 months
  the HbA1c change at 12 months in peers group

SECONDARY OUTCOMES:
Depressive symptoms | 12 months
  the change in the marks of 8-item Patient Health Questionnaire (Chinese version) at 12 months in both peers and peer supporters
Diabetes distress | 12 months
  the change in the marks of Chinese Diabetes Distress Scale (CDDS-15) at 12 months in both peers and peer supporters
Quality of life | 12 months
  the change in the marks of the World Health Organization quality of life questionnaire (WHO-QoL-26) at 12 months in peers and peer supporters
Body weight | 12 months
  the change in body mass index at 12 months in both peers and peer supporters

OTHER OUTCOMES:
Dropout rates of the peer supporters and peers | 12 months
  Dropout rates of the peer supporters and peers
Sustainability of the program | 24 months
  Percentage of peers who still have regular contact with their respective peer supporters after the completion of the program

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Yee-Man Wong, BSc (Nurs), Principal Investigator — HKIDO, CUHK

REFERENCES:
- [Background] Peer Support for Diabetes, Heart Disease and HIV/AIDS: A Review of the Clinical Effectiveness, Cost-effectiveness, and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2013 Nov 8. Available from http://www.ncbi.nlm.nih.gov/books/NBK195174/ PMID 24716255
- [Background] Boothroyd RI, Fisher EB. Peers for progress: promoting peer support for health around the world. Fam Pract. 2010 Jun;27 Suppl 1:i62-8. doi: 10.1093/fampra/cmq017. PMID 20483801
- [Background] Dale JR, Williams SM, Bowyer V. What is the effect of peer support on diabetes outcomes in adults? A systematic review. Diabet Med. 2012 Nov;29(11):1361-77. doi: 10.1111/j.1464-5491.2012.03749.x. PMID 22804713
- [Background] Due-Christensen M, Zoffmann V, Hommel E, Lau M. Can sharing experiences in groups reduce the burden of living with diabetes, regardless of glycaemic control? Diabet Med. 2012 Feb;29(2):251-6. doi: 10.1111/j.1464-5491.2011.03521.x. PMID 22061095
- [Background] Chan JC, Sui Y, Oldenburg B, Zhang Y, Chung HH, Goggins W, Au S, Brown N, Ozaki R, Wong RY, Ko GT, Fisher E; JADE and PEARL Project Team. Effects of telephone-based peer support in patients with type 2 diabetes mellitus receiving integrated care: a randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):972-81. doi: 10.1001/jamainternmed.2014.655. PMID 24781960
- [Background] Zhang Y, Ting R, Lam M, Lam J, Nan H, Yeung R, Yang W, Ji L, Weng J, Wing YK, Sartorius N, Chan JCN. Measuring depressive symptoms using the Patient Health Questionnaire-9 in Hong Kong Chinese subjects with type 2 diabetes. J Affect Disord. 2013 Nov;151(2):660-666. doi: 10.1016/j.jad.2013.07.014. Epub 2013 Jul 31. PMID 23938133